CLINICAL TRIAL: NCT02009852
Title: The Role of microRNA-29b in the Oral Squamous Cell Carcinoma
Acronym: microRNA-29b
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201309076RIN
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Oral Cancer
Keywords: microRNA-29b; Oral squamous cell carcinoma; migration; prognosis
MeSH Terms: conditions — Mouth Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Case-Only
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — tissue, serum, saliva
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Oral cancer: Subjects who suffer from oral cancer.
  Subjects must:
  Should have a blood exam (20ml/each time) before the surgery and 3 months after the surgery.
  In the case the disease recurs after the surgery, subjects need to receive the surgery again and take another blood exam before the surgery and 3 months after the surgery.
  Before the surgery site staff must:
  Collect subjects' saliva once a day (in the morning before breakfast) for 3 consecutive days.
  Collect a 0.5x0.5Cm2 tissue sample of the tumor during the surgery.

SUMMARY:
The Role of microRNA-29b in the Oral Squamous Cell Carcinoma

DETAILED DESCRIPTION:
To find out if there is prognostic value which to the performance of microRNA-29b of oral cancer in Taiwan and provide some reference for future treatment.

We anticipate to enroll 100 persons with oral cancer and collect the tissue which was stained for pathological sections over a 3 year period.

We also collect the blood and saliva samples from patients and the results along with patient-specific information such as tumor phases, tumor size, lymph node metastasis, cancer metastasis, prognosis and betel nut chewing, smoking and drinking habits and other parameters are statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Cancer of the oral cavity.

Exclusion Criteria:

* pregnant woman
* refuse the surgery

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Medical center
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
microRNA-29b | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Shin-Jung Cheng, DDS, MS, PhD, Principal Investigator
Locations (1):
- National Taiwan University Hospital research Ethics Committee, Taipei, Taiwan

REFERENCES:
- [Background] Ambros V. The functions of animal microRNAs. Nature. 2004 Sep 16;431(7006):350-5. doi: 10.1038/nature02871. PMID 15372042
- [Background] Fabbri M, Garzon R, Cimmino A, Liu Z, Zanesi N, Callegari E, Liu S, Alder H, Costinean S, Fernandez-Cymering C, Volinia S, Guler G, Morrison CD, Chan KK, Marcucci G, Calin GA, Huebner K, Croce CM. MicroRNA-29 family reverts aberrant methylation in lung cancer by targeting DNA methyltransferases 3A and 3B. Proc Natl Acad Sci U S A. 2007 Oct 2;104(40):15805-10. doi: 10.1073/pnas.0707628104. Epub 2007 Sep 21. PMID 17890317
- [Background] Pigazzi M, Manara E, Baron E, Basso G. miR-34b targets cyclic AMP-responsive element binding protein in acute myeloid leukemia. Cancer Res. 2009 Mar 15;69(6):2471-8. doi: 10.1158/0008-5472.CAN-08-3404. Epub 2009 Mar 3. PMID 19258499
- [Background] Ma L, Young J, Prabhala H, Pan E, Mestdagh P, Muth D, Teruya-Feldstein J, Reinhardt F, Onder TT, Valastyan S, Westermann F, Speleman F, Vandesompele J, Weinberg RA. miR-9, a MYC/MYCN-activated microRNA, regulates E-cadherin and cancer metastasis. Nat Cell Biol. 2010 Mar;12(3):247-56. doi: 10.1038/ncb2024. Epub 2010 Feb 21. PMID 20173740
- [Background] Ma L, Teruya-Feldstein J, Weinberg RA. Tumour invasion and metastasis initiated by microRNA-10b in breast cancer. Nature. 2007 Oct 11;449(7163):682-8. doi: 10.1038/nature06174. Epub 2007 Sep 26. PMID 17898713
- [Background] Huppi K, Volfovsky N, Mackiewicz M, Runfola T, Jones TL, Martin SE, Stephens R, Caplen NJ. MicroRNAs and genomic instability. Semin Cancer Biol. 2007 Feb;17(1):65-73. doi: 10.1016/j.semcancer.2006.10.004. Epub 2006 Oct 26. PMID 17113784
- [Background] Vokes EE, Weichselbaum RR, Lippman SM, Hong WK. Head and neck cancer. N Engl J Med. 1993 Jan 21;328(3):184-94. doi: 10.1056/NEJM199301213280306. No abstract available. PMID 8417385
- [Background] Fidler IJ. The pathogenesis of cancer metastasis: the 'seed and soil' hypothesis revisited. Nat Rev Cancer. 2003 Jun;3(6):453-8. doi: 10.1038/nrc1098. PMID 12778135
- [Background] Steeg PS. Tumor metastasis: mechanistic insights and clinical challenges. Nat Med. 2006 Aug;12(8):895-904. doi: 10.1038/nm1469. No abstract available. PMID 16892035
- [Background] Gupta GP, Massague J. Cancer metastasis: building a framework. Cell. 2006 Nov 17;127(4):679-95. doi: 10.1016/j.cell.2006.11.001. PMID 17110329
- [Background] Sciume G, Soriani A, Piccoli M, Frati L, Santoni A, Bernardini G. CX3CR1/CX3CL1 axis negatively controls glioma cell invasion and is modulated by transforming growth factor-beta1. Neuro Oncol. 2010 Jul;12(7):701-10. doi: 10.1093/neuonc/nop076. Epub 2010 Feb 8. PMID 20511186
- [Background] Kok SH, Hong CY, Lin SK, Lee JJ, Chiang CP, Kuo MY. Establishment and characterization of a tumorigenic cell line from areca quid and tobacco smoke-associated buccal carcinoma. Oral Oncol. 2007 Aug;43(7):639-47. doi: 10.1016/j.oraloncology.2006.07.007. Epub 2006 Oct 25. PMID 17070096
- [Background] Neville BW, Day TA. Oral cancer and precancerous lesions. CA Cancer J Clin. 2002 Jul-Aug;52(4):195-215. doi: 10.3322/canjclin.52.4.195. PMID 12139232
- [Background] Chang CC, Lin MT, Lin BR, Jeng YM, Chen ST, Chu CY, Chen RJ, Chang KJ, Yang PC, Kuo ML. Effect of connective tissue growth factor on hypoxia-inducible factor 1alpha degradation and tumor angiogenesis. J Natl Cancer Inst. 2006 Jul 19;98(14):984-95. doi: 10.1093/jnci/djj242. PMID 16849681
- [Background] Bartel DP. MicroRNAs: target recognition and regulatory functions. Cell. 2009 Jan 23;136(2):215-33. doi: 10.1016/j.cell.2009.01.002. PMID 19167326
- [Background] Erreni M, Solinas G, Brescia P, Osti D, Zunino F, Colombo P, Destro A, Roncalli M, Mantovani A, Draghi R, Levi D, Rodriguez Y Baena R, Gaetani P, Pelicci G, Allavena P. Human glioblastoma tumours and neural cancer stem cells express the chemokine CX3CL1 and its receptor CX3CR1. Eur J Cancer. 2010 Dec;46(18):3383-92. doi: 10.1016/j.ejca.2010.07.022. Epub 2010 Aug 19. PMID 20728344
- [Background] Gaudin F, Nasreddine S, Donnadieu AC, Emilie D, Combadiere C, Prevot S, Machelon V, Balabanian K. Identification of the chemokine CX3CL1 as a new regulator of malignant cell proliferation in epithelial ovarian cancer. PLoS One. 2011;6(7):e21546. doi: 10.1371/journal.pone.0021546. Epub 2011 Jul 7. PMID 21750716
- [Background] Shiraishi K, Fukuda S, Mori T, Matsuda K, Yamaguchi T, Tanikawa C, Ogawa M, Nakamura Y, Arakawa H. Identification of fractalkine, a CX3C-type chemokine, as a direct target of p53. Cancer Res. 2000 Jul 15;60(14):3722-6. PMID 10919640
- [Background] Moutasim KA, Jenei V, Sapienza K, Marsh D, Weinreb PH, Violette SM, Lewis MP, Marshall JF, Fortune F, Tilakaratne WM, Hart IR, Thomas GJ. Betel-derived alkaloid up-regulates keratinocyte alphavbeta6 integrin expression and promotes oral submucous fibrosis. J Pathol. 2011 Feb;223(3):366-77. doi: 10.1002/path.2786. Epub 2010 Oct 25. PMID 21171082
- [Background] Thiery JP, Acloque H, Huang RY, Nieto MA. Epithelial-mesenchymal transitions in development and disease. Cell. 2009 Nov 25;139(5):871-90. doi: 10.1016/j.cell.2009.11.007. PMID 19945376